CLINICAL TRIAL: NCT00229658
Title: A Prospective, Open-Label, Observational Study Evaluating SYMLIN® (Pramlintide Acetate) Injection Use in Insulin Using Patients With Type 2 and Type 1 Diabetes Following SYMLIN Introduction Into the Marketplace
Brief Title: An Observational Study Evaluating SYMLIN® (Pramlintide Acetate) Injection Use in Insulin Using Patients With Type 2 and Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 137-161
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Results first posted 2009-06-24 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-02

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: diabetes; pramlintide; Symlin; Amylin; phase 4
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — pramlintide

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1: Patients with type 1 diabetes
  Interventions: Drug: pramlintide acetate
- Type 2: Patients with type 2 diabetes
  Interventions: Drug: pramlintide acetate

INTERVENTIONS:
Drug: pramlintide acetate — Subcutaneous injection prior to each major meal
  Other Names: Symlin

SUMMARY:
This is an open label, observational study designed to collect data that characterize the use of SYMLIN following the introduction of the medication into the marketplace. Health care providers and subjects selected for study participation are intended to be representative of those providers prescribing, and subjects receiving, SYMLIN therapy.

ELIGIBILITY:
Inclusion Criteria:

* The following inclusion criteria are consistent with information in the SYMLIN package insert and apply to insulin using patients with type 2 or type 1 diabetes who:

  * Have failed to achieve the desired or optimal level of glycemic control despite utilizing appropriate, individualized insulin regimens
  * Have A1C <=9.0% within 3 months of study enrollment
  * Are receiving ongoing diabetes care under the guidance of a Health Care Provider (HCP) trained in the use of SYMLIN

Exclusion Criteria:

* The following exclusion criteria are consistent with the SYMLIN package insert and specifically exclude patients who:

  * Are poorly compliant with their current insulin regimen, as defined by their HCP
  * Are poorly compliant with prescribed blood glucose self monitoring, as defined by their HCP
  * Have experienced recurrent patient-ascertained severe hypoglycemia requiring assistance during the past 6 months
  * Have hypoglycemia unawareness
  * Have a confirmed diagnosis of gastroparesis
  * Require the use of drugs that stimulate gastrointestinal motility
  * Are female and pregnant or lactating and for whom the HCP determines the potential benefit does not justify the potential risk to the fetus or infant
  * Have been treated with SYMLIN within 3 months prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cross-section of clinical practice settings
Sampling Method: Non-Probability Sample
Enrollment: 1297 (Actual)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Medical Development, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (107):
- United States (107):
  - Research Site, Birmingham, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Encinitas, California
  - Research Site, Escondido, California
  - Research Site, Fresno, California
  - Research Site, Lafayette, California
  - Research Site, Moreno Valley, California
  - Research Site, Sacramento, California
  - Research Site, Salinas, California
  - Research Site, Santa Barbara, California
  - Research Site, Torrance, California
  - Research Site, Vacaville, California
  - Research Site, Arvada, Colorado
  - Research Site, Aurora, Colorado
  - Research Site, Norwalk, Connecticut
  - Research Site, Wilmington, Delaware
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Maitland, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Plantation, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Canton, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Valdosta, Georgia
  - Research Site, ‘Aiea, Hawaii
  - Research Site, Caldwell, Idaho
  - Research Site, Idaho Falls, Idaho
  - Research Site, Pocatello, Idaho
  - Research Site, Evergreen Park, Illinois
  - Research Site, Wheaton, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Franklin, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Shawnee Mission, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Laplace, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Bloomfield, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Eagan, Minnesota
  - Research Site, Butte, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Hamilton, New Jersey
  - Research Site, Jersey City, New Jersey
  - Research Site, Livingston, New Jersey
  - Research Site, Moorestown, New Jersey
  - Research Site, Neptune City, New Jersey
  - Research Site, North Plainfield, New Jersey
  - Research Site, Albany, New York
  - Research Site, Binghamton, New York
  - Research Site, Forest Hills, New York
  - Research Site, Lawrence, New York
  - Research Site, New York, New York
  - Research Site, Riverhead, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, Utica, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Mentor, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Bridgeville, Pennsylvania
  - Research Site, Carlisle, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Sewickley, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Sumter, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Hendersonville, Tennessee
  - Research Site, Hixon, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Provo, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, McLean, Virginia
  - Research Site, Norton, Virginia
  - Research Site, Puyallup, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Walla Walla, Washington
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Pencek R, Roddy T, Peters Y, De Young MB, Herrmann K, Meller L, Nguyen H, Chen S, Lutz K. Safety of pramlintide added to mealtime insulin in patients with type 1 or type 2 diabetes: a large observational study. Diabetes Obes Metab. 2010 Jun;12(6):548-51. doi: 10.1111/j.1463-1326.2010.01201.x. PMID 20518811

RESULTS

PARTICIPANT FLOW:
Groups:
- Type 1 Diabetes: Insulin using patients with Type 1 diabetes
- Type 2 Diabetes: Insulin using patients with Type 2 diabetes
Period: Overall Study
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Started | 766 | 531
Completed | 541 | 364
Not Completed | 225 | 167
Not completed — Administrative | 2 | 1
Not completed — Investigator decision | 13 | 10
Not completed — Other | 80 | 60
Not completed — Lost to Follow-up | 82 | 55
Not completed — Serious Adverse Event | 2 | 2
Not completed — Withdrawal of consent | 46 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 1 Diabetes | Type 2 Diabetes | Total
Number analyzed (Participants) | 766 | 531 | 1297
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 0 | 8
  Between 18 and 65 years | 721 | 406 | 1127
  >=65 years | 37 | 125 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.22) | 56.9 (11.10) | 48.8 (14.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 500 | 296 | 796
  Male | 266 | 235 | 501
Region of Enrollment [Number; unit: participants]
  United States | 766 | 531 | 1297
Body Weight [Mean (Standard Deviation); unit: kg] | 87.21 (19.843) | 112.53 (24.790) | 97.57 (25.273)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 20.66 (11.709) | 14.76 (8.355) | 18.24 (10.857)
HbA1c [Mean (Standard Deviation); unit: %] | 7.86 (1.082) | 8.23 (1.538) | 8.01 (1.301)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Patient-Ascertained Severe Hypoglycemia (PASH) During the Adjustment Period
Description: PASH is defined as episodes of hypoglycemia requiring the assistance of another individual (including aid in ingestion of oral carbohydrate); and/or requiring the administration of glucagon injection, intravenous glucose, or other medical intervention. The adjustment period represents the initial 0-3 months of pramlintide treatment
Time Frame: 0-3 months
Population: Intent-to-Treat
Measure: Number; unit: Incidence (%)
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 766 | 531
Incidence (%) | 4.8 | 2.8

2. Primary Outcome: Annual Event Rate of Patient-Ascertained Severe Hypoglycemia (PASH) During the Adjustment Period
Description: The annual event rate was calculated as the total number of events during the time period divided by the total years of exposure to pramlintide for all patients during the time period. The adjustment period represents the initial 0-3 months of pramlintide treatment.
  PASH is defined as episodes of hypoglycemia requiring the assistance of another individual (including aid in ingestion of oral carbohydrate); and/or requiring the administration of glucagon injection, intravenous glucose, or other medical intervention.
Time Frame: 0-3 months
Population: Intent-to-Treat
Measure: Number; unit: Events per patient year
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 766 | 531
Events per patient year | 0.3255 | 0.1941

3. Secondary Outcome: The Incidence of Patient-Ascertained Severe Hypoglycemia (PASH) During the Steady State Period
Description: The steady state period represents the >3-6 months of pramlintide treatment following the adjustment period.
  PASH is defined as episodes of hypoglycemia requiring the assistance of another individual (including aid in ingestion of oral carbohydrate); and/or requiring the administration of glucagon injection, intravenous glucose, or other medical intervention.
Time Frame: >3-6 months
Population: Intent-to-Treat, number analyzed includes patients still enrolled in the study during the steady-state period (3-6 months)
Measure: Number; unit: Incidence (%)
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 512 | 387
Incidence (%) | 1.8 | 0.3

4. Secondary Outcome: The Annual Event Rate of Patient-Ascertained Severe Hypoglycemia (PASH) During the Steady State Period
Description: The annual event rate was calculated as the total number of events during the time period divided by the total years of exposure to pramlintide for all patients during the time period. The steady state period represents the >3-6 months of pramlintide treatment following the adjustment period.
  PASH is defined as episodes of hypoglycemia requiring the assistance of another individual (including aid in ingestion of oral carbohydrate); and/or requiring the administration of glucagon injection, intravenous glucose, or other medical intervention.
Time Frame: >3-6 months
Population: as for outcome 3
Measure: Number; unit: Events per patient year
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 512 | 387
Events per patient year | 0.0844 | 0.0248

5. Secondary Outcome: Incidence of Medically Assisted Severe Hypoglycemia (MASH) During the Adjustment Period
Description: MASH is defined as episodes of severe hypoglycemia requiring IM glucagon, IV glucose, hospitalization, paramedic assistance, emergency room visit, and/or is assessed as a serious adverse event (SAE) by the investigator. MASH is a subset of PASH. The adjustment period represents the initial 0-3 months of pramlintide treatment
Time Frame: 0-3 months
Population: Intent-to-Treat.
Measure: Number; unit: Incidence (%)
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 766 | 531
Incidence (%) | 1.8 | 0.4

6. Secondary Outcome: The Annual Event Rate of Medically Assisted Severe Hypoglycemia (MASH) During the Adjustment Period
Description: The annual event rate was calculated as the total number of events during the time period divided by the total years of exposure to pramlintide for all patients during the time period. The adjustment period represents the initial 0-3 months of pramlintide treatment.
  MASH is defined as episodes of severe hypoglycemia requiring IM glucagon, IV glucose, hospitalization, paramedic assistance, emergency room visit, and/or is assessed as a serious adverse event (SAE) by the investigator. MASH is a subset of PASH.
Time Frame: 0-3 months
Population: Intent-to-Treat
Measure: Number; unit: Events per patient year
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 766 | 531
Events per patient year | 0.0996 | 0.0185

7. Secondary Outcome: Incidence of Medically Assisted Severe Hypoglycemia (MASH) During the Steady State Period
Description: The steady state period represents the >3-6 months of pramlintide treatment following the adjustment period.
  MASH is defined as episodes of severe hypoglycemia requiring IM glucagon, IV glucose, hospitalization, paramedic assistance, emergency room visit, and/or is assessed as a serious adverse event (SAE) by the investigator. MASH is a subset of PASH.
Time Frame: >3-6 months
Population: as for outcome 3
Measure: Number; unit: Incidence (%)
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 512 | 387
Incidence (%) | 0.8 | 0.3

8. Secondary Outcome: Annual Event Rate of Medically Assisted Severe Hypoglycemia (MASH) During the Steady State Period
Description: The annual event rate was calculated as the total number of events during the time period divided by the total years of exposure to pramlintide for all patients during the time period. The steady state period represents the >3-6 months of pramlintide treatment following the adjustment period.
  MASH is defined as episodes of severe hypoglycemia requiring IM glucagon, IV glucose, hospitalization, paramedic assistance, emergency room visit, and/or is assessed as a serious adverse event (SAE) by the investigator. MASH is a subset of PASH.
Time Frame: >3-6 months
Population: as for outcome 3
Measure: Number; unit: Events per patient year
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 512 | 387
Events per patient year | 0.0375 | 0.0124

9. Secondary Outcome: Change in HbA1c From Baseline at Month 3
Description: Change in HbA1c from baseline at month 3. The HbA1c test measures the percent of glycosylated hemoglobin in the blood.
Time Frame: 3 months
Population: Intent-to-Treat, patients who discontinue SYMLIN 7 or more days prior to a site visit are not included in the analyses
Measure: Mean (Standard Error); unit: percent
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 414 | 371
percent | -0.12 (0.037) | -0.33 (0.056)

10. Secondary Outcome: Change in HbA1c From Baseline at Month 6
Description: Change in HbA1c from baseline at month 6. The HbA1c test measures the percent of glycosylated hemoglobin in the blood.
Time Frame: 6 months
Population: Intent-to-Treat, patients who discontinue SYMLIN 7 or more days prior to a site visit are not included in the analyses
Measure: Mean (Standard Error); unit: percent
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 347 | 290
percent | -0.26 (0.046) | -0.44 (0.071)

11. Secondary Outcome: Change in Body Weight From Baseline at Month 3
Description: Mean change in body weight from baseline at month 3
Time Frame: 3 months
Population: Intent-to-Treat, patients who discontinue SYMLIN 7 or more days prior to a site visit are not included in the analyses
Measure: Mean (Standard Error); unit: kg
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 443 | 370
kg | -1.95 (0.154) | -1.94 (0.237)

12. Secondary Outcome: Change in Body Weight From Baseline at Month 6
Description: Mean change in body weight from baseline at month 6
Time Frame: 6 months
Population: Intent-to-Treat, patients who discontinue SYMLIN 7 or more days prior to a site visit are not included in the analyses
Measure: Mean (Standard Error); unit: kg
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 364 | 294
kg | -2.77 (0.246) | -1.98 (0.322)

ADVERSE EVENTS:
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Serious Adverse Events (participants affected / at risk) | 14 | 13
Other Adverse Events (participants affected / at risk) | 0/766 | 0/531
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Type 1 Diabetes | Type 2 Diabetes
Angina pectoris (Cardiac disorders) | 1/766 | 0/531
Angina unstable (Cardiac disorders) | 1/766 | 0/531
Atrioventricular block complete (Cardiac disorders) | 0/766 | 1/531
Cardiac failure congestive (Cardiac disorders) | 1/766 | 1/531
Coronary artery disease (Cardiac disorders) | 0/766 | 1/531
Myocardial infarction (Cardiac disorders) | 0/766 | 1/531
Pancreatitis (Gastrointestinal disorders) | 1/766 | 0/531
Chest pain (General disorders) | 0/766 | 1/531
Hernia obstructive (General disorders) | 0/766 | 1/531
Cholecystitis acute (Hepatobiliary disorders) | 1/766 | 0/531
Appendicitis (Infections and infestations) | 1/766 | 0/531
Cellulitis (Infections and infestations) | 0/766 | 1/531
Diverticulitis (Infections and infestations) | 0/766 | 1/531
Osteomyelitis (Infections and infestations) | 0/766 | 1/531
Pneumonia (Infections and infestations) | 1/766 | 0/531
Sepsis (Infections and infestations) | 0/766 | 2/531
Urosepsis (Infections and infestations) | 0/766 | 1/531
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3/766 | 0/531
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1/766 | 0/531
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/766 | 0/531
Ovarian granulosa-theca cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/766 | 1/531
Presyncope (Nervous system disorders) | 1/766 | 0/531
Syncope (Nervous system disorders) | 1/766 | 0/531
Ureteric stenosis (Renal and urinary disorders) | 0/766 | 1/531
Ovarian cyst (Reproductive system and breast disorders) | 1/766 | 0/531
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/766 | 1/531
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/766 | 1/531
Skin ulcer (Skin and subcutaneous tissue disorders) | 0/766 | 1/531
Deep vein thrombosis (Vascular disorders) | 1/766 | 0/531

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less